CLINICAL TRIAL: NCT01639690
Title: A Phase I Clinical Trial for the Treatment of ß-Thalassemia Major with Autologous CD34+ Hematopoietic Progenitor Cells Transduced with TNS9.3.55 a Lentiviral Vector Encoding the Normal Human ß-Globin Gene
Brief Title: ß-Thalassemia Major with Autologous CD34+ Hematopoietic Progenitor Cells Transduced with TNS9.3.55 a Lentiviral Vector Encoding the Normal Human ß-Globin Gene
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: San Rocco Therapeutics (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-164
Record Dates: First submitted 2012-07-11; First posted 2012-07-13 (Estimated); Last update posted 2024-10-16 (Actual); Status verified 2024-09

CONDITIONS: Confirmed Diagnosis of ß-thalassemia Major
Keywords: BUSULFAN; G-CSF; CliniMACS-CD34 Reagent System; Blood transfusion; 10-164; Autologous CD34+ cells transduced with TNS9.3.55, a lentiviral vector encoding the human β-globin gene
MeSH Terms: interventions — Blood Component Removal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Autologous CD34+ cells transduced with TNS9.3.55 (Experimental): An open label study using a non-myeloablative conditioning regimen of busulfan and 1 or several infusions of autologous hematopoietic stem cells transduced with a lentiviral vector encoding the human ß-globin gene.
  Interventions: Genetic: Autologous CD34+ cells transduced with TNS9.3.55

INTERVENTIONS:
Genetic: Autologous CD34+ cells transduced with TNS9.3.55 — Patients will receive Filgrastim followed by apheresis of peripheral blood stem cells. CD34+ cells will be purified and transduced ex vivo. Transduced cells will be frozen in several aliquots whenever possible while vector copy number determination and biosafety testing are performed. Patients will be treated in the outpatient and/or inpatient units, and receive intravenous busulfan (8mg/kg) as non-myeloablative conditioning. Patients will be administered 2-12 x 10^6 transduced CD34+ cells per kg in 1 or several infusions. A back-up of 2 x 10^6 untransduced CD34+ cells per kg will be preserved for every patient.
  Other Names: Patient treatment with Filgrastim will last for up to 6 days with apheresis; collection on days 4 and 5 or days 5 or 6 if required. Reduced Intensity Conditioning will; consist of two days of busulfan treatment with an interval of two days prior to transplantation.; Intravenous infusion of autologous CD34+ cells transduced with TNS9.3.55 will; be administered over 15-30 minutes in a volume of approximately 50 to 250 mL; on day 0. Subsequent infusions of autologous CD34+ cells transduced with TNS9.3.55; may be administered on day +1 or thereafter.

SUMMARY:
The patient has inherited ß-thalassemia major through the genes. These genes have mistakes in them, so the body cannot make normal red blood cells. Stem cells are made in the bone marrow. They are the earliest form of blood cells.

This study is being done to see if the investigators can make the stem cells produce normal red blood cells and hemoglobin. The investigators do this by collecting the stem cells. The genes with mistakes are removed from the cells. These cells are then treated so they have the corrected gene for making normal hemoglobin. These treated cells are given back to the patient through an injection (shot) in the vein. This is also known as gene transfer. In order for the body to accept these cells, the patient will need to receive a low dose of a drug called busulfan. It is a drug that will prepare the body to receive the new stem cells.

This study will let the investigators know:

* If it is safe to give the patient the treated stem cells
* If the treated stem cells will go into the bone marrow without causing side effects.

Gene transfer has been used for the past five years. It has been successful in treating many blood disorders. At least 20 patients have received the type of treatment that the patient will get on this study. This treatment for B-thalassemia major was developed at Memorial Sloan Kettering (MSK). It was studied for a long time in the lab before being given to patients.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be 18 years or older
* Subjects may be of either gender or of any ethnic background
* Subjects must have a confirmed diagnosis of ß-thalassemia major and have been enrolled in a hypertransfusion program with a confirmed annual transfusion of ≥100 mL/kg/yr but < 200 mL/kg/yr, AND ≥ 8 transfusions of blood per year over a minimum of two years.
* Patients must NOT have an HLA-matched sibling
* Patients must be off hydroxyurea (HU) or erythropoietin (EPO) treatment for at least three months prior to entry onto the study
* Subjects must have a performance score of Karnofsky ≥70% at the time of entry into the study.
* Subjects must have liver iron value of < 15 mg/g/dry weight Iron quantitation may be performed by imaging such as T2*MRI or by biopsy
* Subjects must have no evidence of cirrhosis** of the liver. Fibrosis of the liver can be tested by Fibroscan (47, 48, 49), or by liver biopsy. These should be performed within approximately a one year period prior to entry onto the study.
* Subjects with an evaluation of cardiac function indicating:
* normal function on MUGA scan (Multiple Gated Acquisition scan) or other methodology.

And

* Patients must have a left ventricular ejection fraction (LVEF) of ≥ 60% and/or T2*MRI cardiac evaluation with T2* ≥20 milliseconds
* Subjects with asymptomatic pulmonary function based on Lung Diffusion Testing DLCO Test DLCO ≥ 50% of predicted (corrected for hemoglobin)
* Subjects with a determination of renal function based on: serum creatinine < than or = to 1.5 mg/dL or if serum creatinine is outside the normal range, then CrCl > 60-ml/min/1.73 m2
* Subjects must have adequate hepatic function based on:
* < 3 x ULN ALT and
* < 2.0 total serum bilirubin (unless secondary to hemolysis)
* Patients must be available for follow-up evaluations at 30, 60, 180 days post BMT and yearly thereafter indefinitely.

  * The possibility of unrelated donor stem cell transplantation will be discussed with patients, and a "preliminary" search for an unrelated donor may be done at the request of the patient. However, the finding of a potential HLA-matched unrelated donor will not exclude the patient from participating into this trial).

    * As the inclusion criteria are more specific than the Lucarelli/Pesaro thalassemia pre-transplant classification (Class 1,2 or 3 according to presence or absence of fibrosis, adequate chelation and/or hepatomegaly), the criteria stated above will be used in lieu of the Lucarelli/Pesaro classification.

Exclusion Criteria:

* Active infections including Hepatitis B and Hepatitis C***,
* Active infections including HTLV 1 and 2, and HIV 1 and 2
* Patients with treated HLTV or HIV
* Diabetes Mellitus
* Bone Marrow myelodysplasia and/or chromosomal abnormalities
* Female patient pregnant or breast feeding
* Patients with uncontrolled seizure disorders
* Patients with severe pulmonary hypertension Tricuspid Jet velocity > 2.5 m/sec
* Family history of familial cancer syndromes (leukemia, breast, ovarian, colorectal, etc.)

  *** Definition of active Hepatitis C include:
* Positive HCV RNA Viral load by quantitative PCR testing Or if Negative HCV RNA viral load BUT on antiviral treatment
* Liver biopsy with pathologic evidence of
* Necrosis and inflammation around the portal areas - piecemeal necrosis or interface hepatitis or necrosis of hepatocytes and focal inflammation in the liver parenchyma.
* Inflammatory cells in the portal areas ("portal inflammation").
* Fibrosis, with early stages being confined to the portal tracts, intermediate stages being expansion of the portal tracts and bridging between portal areas or to the central area, and late stages being frank cirrhosis characterized by architectural disruption of the liver with fibrosis and regeneration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2012-07; Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
safety | 2 years
  of transplanted autologous CD34+ hematopoietic cells that are transduced ex vivo with TNS9.3.55 and transplanted in subjects with ß-thalassemia major conditioned with a reduced-intensity non-myeloablative preparative regimen.
  1. The occurrence of insertional oncogenesis, which will be investigated by monitoring peripheral blood cell counts and leukocyte clonality using FACS analysis, qPCR for vector. copy number, LAM-PCR and/or 454 sequencing;
  2. The generation of a replication-competent lentivirus (RCL).
  3. The safety of a low dose non-myeloablative conditioning regimen
tolerability | 2 years
  of transplanted autologous CD34+ hematopoietic cells that are transduced ex vivo with TNS9.3.55 & transplanted in subjects with ß-thalassemia major conditioned with a reduced-intensity non-myeloablative preparative regimen. monitoring the following: 1. The occurrence of insertional oncogenesis, which will be investigated by monitoring peripheral blood cell counts & leukocyte clonality using FACS analysis, qPCR for vector. copy number, LAM-PCR and/or 454 sequencing; 2.The generation of a replication-competent lentivirus (RCL). 3.The safety of a low dose non-myeloablative conditioning regimen

SECONDARY OUTCOMES:
the level of engraftment | 2 years
  of the genetically modified autologous CD34+ cells and expression of the transduced ß-globin gene as measured by: Blood for measurement of vector copy number and transgene expression in blood cells at months 1, 2 and 3.
  - Bone Marrow Samples for evaluation of CFU, BFU-E gene+ colonies and Q-PCR will be tested at month 1.
The frequency of post transplant palliative transfusions | 2 years
  The number of red blood cell transfusions after engraftment will be quantitatively evaluated for efficacy purposes.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital "V.Cervello" Uoc Ematologiaii E Malattie Rare, Palermo, Italy

REFERENCES:
- [Derived] Boulad F, Maggio A, Wang X, Moi P, Acuto S, Kogel F, Takpradit C, Prockop S, Mansilla-Soto J, Cabriolu A, Odak A, Qu J, Thummar K, Du F, Shen L, Raso S, Barone R, Di Maggio R, Pitrolo L, Giambona A, Mingoia M, Everett JK, Hokama P, Roche AM, Cantu VA, Adhikari H, Reddy S, Bouhassira E, Mohandas N, Bushman FD, Riviere I, Sadelain M. Lentiviral globin gene therapy with reduced-intensity conditioning in adults with beta-thalassemia: a phase 1 trial. Nat Med. 2022 Jan;28(1):63-70. doi: 10.1038/s41591-021-01554-9. Epub 2022 Jan 3. PMID 34980909
- [Derived] Boulad F, Wang X, Qu J, Taylor C, Ferro L, Karponi G, Bartido S, Giardina P, Heller G, Prockop SE, Maggio A, Sadelain M, Riviere I. Safe mobilization of CD34+ cells in adults with beta-thalassemia and validation of effective globin gene transfer for clinical investigation. Blood. 2014 Mar 6;123(10):1483-6. doi: 10.1182/blood-2013-06-507178. Epub 2014 Jan 15. PMID 24429337
- See also: San Rocco Therapeutics — https://sanroccotherapeutics.com/